CLINICAL TRIAL: NCT03657901
Title: Sleep, Stress and Learning: an Experimental Pilot Study
Acronym: Sleepstress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anu-Katriina Pesonen, Professor, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Sleepstress
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Stress; Sleep

STUDY DESIGN:
Intervention Model Description: Randomized control trial with a cross-over design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing (Experimental): Guided slow breathing for 30 minutes before sleep onset
  Interventions: Behavioral: Slow breathing
- Music listening (Active Comparator): Guided music listening for 30 minutes before sleep onset
  Interventions: Behavioral: Music listening

INTERVENTIONS:
Behavioral: Music listening — Guided music listening for 30 minutes before sleep onset
  Arms: Music listening
Behavioral: Slow breathing — Guided slow breathing for 30 minutes before sleep onset
  Arms: Breathing

SUMMARY:
To investigate the efficiency and effect of a programmed slow-breathing exercise in the evening to the heart rate variability, sleep quality and memory performance over night.

DETAILED DESCRIPTION:
Background Stress and increased alertness in the evening are major reasons for sleep onset problems, poor sleep and insomnia symptoms. For instance, increased amount of REM, and decreased amount of slow wave sleep may result. Also, the function of sleep in memory consolidation may suffer. They also affect the sleep structure and continuity during the night. They are highly prevalent phenomena among the entire population, including healthy adults and children. However, at the physiological level, the concept of evening alertness is still understudied and often neglected.

Recent advances show that breathing exercise is an efficient tool to reduce stress. However, its use specifically prior to sleep onset and with measurement sleep stages and their microstructures with sleep EEG has been little been studied before. The overall objective of this study is to explore interrelations of stress, learning and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* age 20-45

Exclusion Criteria:

* chronic disease requiring daily medication, acute sickness (e.g. a flu), jet lag from a recent travel, current diagnosed sleep disorder (such as snoring or insomnia) and any use of medication affecting autonomic nervous system function or sleep.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 10 males, 10 females
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep structure | Change from night 1 to night 2
  Percent distribution of different sleep stages

SECONDARY OUTCOMES:
Sleep spindle duration | Change from night 1 to night 2
  Duration of sleep spindles in seconds
Sleep spindle power | Change from night 1 to night 2
  Amplitude of sleep spindles in microvolts

CONTACTS AND LOCATIONS:
Overall Officials: Anu-Katriina Pesonen, prof, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sleep lab home page — https://www.helsinki.fi/en/researchgroups/sleep-and-mind